CLINICAL TRIAL: NCT05466747
Title: Randomized, Open-label, Parallel-group, Multicenter, Non-inferiority and Dose-response Study to Evaluate the Efficacy and Safety of RYMPHYSIA (ARALAST NP) for Alpha1-Proteinase Inhibitor (A1PI) Augmentation Therapy in Subjects With A1PI Deficiency and Chronic Obstructive Pulmonary Disease-Emphysema
Brief Title: A Study of RYMPHYSIA for Alpha1-Proteinase Inhibitor (A1PI) Therapy in Adults With A1PI Deficiency and Chronic Obstructive Pulmonary Disease (COPD)-Emphysema
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-883-4002; 2022-502171-30-00 (Other: EU CTIS)
Record Dates: First submitted 2022-06-17; First posted 2022-07-20 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Alpha1-Antitrypsin Deficiency
Keywords: TAK-883; Chronic Obstructive Pulmonary Disease; RYMPHYSIA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: RYMPHYSIA 60 mg/kg (Experimental): Participants will receive 60 mg/kg RYMPHYSIA, intravenous (IV) infusion, once every week for up to 104 weeks.
  Interventions: Biological: RYMPHYSIA
- Part A: Another Available A1PI 60 mg/kg (Active Comparator): Participants will receive 60 mg/kg of another available A1PI, IV infusion, once every week for up to 104 weeks.
  Interventions: Biological: Another Available A1PI
- Part B: RYMPHYSIA 60 mg/kg (Experimental): Participants will receive 60 mg/kg RYMPHYSIA, IV infusion, once every week for up to 104 weeks.
  Interventions: Biological: RYMPHYSIA
- Part B: RYMPHYSIA 120 mg/kg (Experimental): Participants will receive 120 mg/kg RYMPHYSIA, IV infusion, once every week for up to 104 weeks.
  Interventions: Biological: RYMPHYSIA

INTERVENTIONS:
Biological: RYMPHYSIA — RYMPHYSIA administered through an IV injection.
  Other Names: Alpha1-PI; TAK-883; A1PI; Alpha1-Proteinase Inhibitor (Human); ARALAST NP
  Arms: Part A: RYMPHYSIA 60 mg/kg; Part B: RYMPHYSIA 120 mg/kg; Part B: RYMPHYSIA 60 mg/kg
Biological: Another Available A1PI — Another available A1PI administered through an IV injection.
  Other Names: Alpha1-PI; Alpha1-Proteinase Inhibitor (Human)
  Arms: Part A: Another Available A1PI 60 mg/kg

SUMMARY:
The main purpose of this study is to evaluate the efficacy of RYMPHYSIA [Alpha1-Proteinase Inhibitor (Human)] compared to another available alpha-1 proteinase Inhibitor (A1PI) in adults with A1PI deficiency and COPD-emphysema.

In Part A of the study, participants will be randomly assigned to receive either RYMPHYSIA or another available A1PI for 104 weeks. Participants who were randomized to another available A1PI will enter a 2-week follow-up period after the treatment phase is completed; participants who were randomized to RYMPHYSIA will enter Part B.

In Part B, participants will be randomly assigned to one of two groups and will receive either the same dose of RYMPHYSIA as in Part A or a different dose for an additional 104 weeks, followed by a 2-week follow-up period.

ELIGIBILITY:
Inclusion:

* Adult 18 to 75 years at the time of screening.
* Diagnosis of alpha1-proteinase inhibitor (A1PI) deficiency, defined as follows:

  * Endogenous serum A1PI level lesser than (<)11 micromolar (μM) or 57.2 micrograms per deciliter (mg/dL) (0.572 gram per liter [g/L]) (as measured at the end of the washout, if applicable)
  * Genotype ZZ, Z/null, null/null, MMalton/Z, or others that result in A1PI levels <11 μM. Prior documentation of genotype will be sufficient, or genotyping will be offered at the time of screening
* Participants eligible for enrollment include newly diagnosed, previously untreated, currently treated, and currently not on treatment but who have received treatment in the past. For those currently on augmentation therapy, a 2-week minimum washout is required until A1PI levels are <11 μM.
* Clinically evident chronic obstructive pulmonary disease (COPD)-emphysema at the time of screening defined by post-bronchodilator FEV1 of greater than or equal to (≥)30 percent (%) and lesser than or equal to (≤)80% predicted and FEV1/forced vital capacity (FVC) <70%, corresponding to mild to severe COPD (according to Global Initiative for Chronic Obstructive Lung Disease [GOLD] Criteria, stage I-III) (Global Initiative for Chronic Obstructive Lung Disease 2021) and evidence of emphysema on chest imaging (confirmed by the baseline computer topography [CT] densitometry scan).
* If treated with any respiratory medications including inhaled bronchodilators, inhaled corticosteroids, or systemic corticosteroids (e.g., prednisone ≤10 micrograms per day [mg/day] or its equivalent), the doses of medications should have remained stable for at least 28 days prior to screening.
* No clinically significant abnormalities (other than emphysema, bronchitis, or bronchiectasis) detected via chest imaging at the time of screening.
* Males and non-pregnant, non-lactating females whose screening pregnancy test is negative and willing and able to employ adequate contraceptive methods.
* Willing and able to refrain from smoking (including e-cigarettes and vaping of any other substance) for the duration of study.
* Willing and able to comply with the requirements of the protocol and able to voluntarily provide written, signed, and dated (personally or via a legally authorized representative) informed consent to participate in the study.

Exclusion:

* Known ongoing or history of clinically significant disease other than respiratory or liver disease secondary to A1PI deficiency.
* If experiencing COVID-19, lower respiratory tract infection (LRTI) and/or acute COPD exacerbation at the time of screening. Participants may be re-screened after clinical resolution of COVID-19, LRTI and/or acute COPD exacerbation and must have also remained stable for at least 6 weeks after the onset of illness.
* Known ongoing or history of clinically significant cor pulmonale and/or congestive heart failure with New York Heart Association (NYHA) Class III/IV symptoms.
* Has received an organ transplant, has undergone major lung surgery (e.g., lung volume reduction surgery or lobectomy surgery), or is currently on a transplant waiting list.
* Experiencing an active malignancy or has a history of malignancy within 5 years prior to screening, with the exception of the following: adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or stable prostate cancer not requiring treatment.
* Current active smoker (including e-cigarettes or vaping, nicotine or any other substance). A participant with a previous history of smoking has to have ceased active smoking at least 6 months prior to screening. Participants with a positive nicotine/cotinine test due to nicotine replacement therapy (eg, patches, chewing gum) or snuff are eligible.
* Receiving long-term therapy (>28 days) of parenteral corticosteroids or oral corticosteroids at doses greater than 10 mg/day of prednisone or its equivalent.
* Receiving chronic 24 hours/day oxygen supplementation (other than for an acute COPD exacerbation, or supplemental oxygen with continuous positive airway pressure [CPAP], or bi-level positive airway pressure [BiPAP] for acute respiratory failure).
* Known selective immunoglobulin A (IgA) deficiency (IgA level <7 mg/dL at screening) with anti-IgA antibodies and a history of any hypersensitivity reaction.
* Known history of hypersensitivity following infusions of human immunoglobulins, human albumin, blood or blood components.
* Presence of clinically significant laboratory abnormalities at the screening that in the opinion of the investigator would impact the participant's safety if enrolled in the study.
* Presence of any of the following that, in the opinion of the investigator, would affect participant's safety or compliance or confound the results of the study, including known clinically significant medical, psychiatric, or cognitive illness, is a recreational drug/alcohol user, or has any other uncontrolled medical condition (e.g., unstable angina, transient ischemic attack, uncontrolled hypertension).
* Known exposure to another investigational product/investigational medicinal product (IP/IMP) within 28 days prior to enrollment or is scheduled to participate in another clinical study involving an IP/IMP or investigational device during this study.
* Participant is a family member or employee of the investigator.
* If female, participant is pregnant or nursing at the time of enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-04-26 (Estimated); Study Completion 2029-05-07 (Estimated)

PRIMARY OUTCOMES:
Part A: Annual Rate of Change in the Physiologically Adjusted Lung Density | Up to Week 104
  Annual rate of the physiologically adjusted lung density change will be measured as the 15th percentile (PD15) of the lung density measurements as assessed by computed tomography (CT) densitometry at total lung capacity (TLC). CT lung density at the 15th percentile (PD15) is the threshold below which 15 percent (%) of the voxels have lower densities and is used as the parameter for estimating the rate of lung density decline.

SECONDARY OUTCOMES:
Part A: Annual Rate of Change in the Plasma Level of Elastin Degradation Products | Up to Week 104
  The annual rate of change in the plasma levels of elastin degradation products (desmosine and isodesmosine) will be assessed to document the pharmacodynamic (PD) effect of RYMPHYSIA on the activity of neutrophil elastase using high-performance liquid chromatography-mass spectrometry (LC-MS). The assessment of elastin degradation products will be performed for participants in the RYMPHYSIA treatment arm only.
Part A: Annual Rate of Change in the Plasma Level of Fibrinogen Degradation Products | Up to Week 104
  The annual rate of change in the plasma levels of fibrinogen degradation products (Aα-Val360 fragments) will be assessed to document the PD effect of RYMPHYSIA on the activity of neutrophil elastase using high-performance LC-MS. The assessment of fibrinogen degradation products will be performed for participants in the RYMPHYSIA treatment arm only.
Part A and Part B: Number of Moderate or Severe Exacerbations of Chronic Obstructive Pulmonary Disease (COPD) | Part A, Part B: Up to Week 104
  COPD exacerbations are defined as an acute worsening of respiratory symptoms that results in additional therapy and will be assessed based on the classification in GOLD criteria (2021). The assessment of COPD exacerbations will be performed for participants in the RYMPHYSIA treatment arm only.
Part A and Part B: Annual Rate of Change in the Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) | Part A, Part B: Up to Week 104
  FEV1 is the volume of air that can be forcefully exhaled in the first second after a full inspiration obtained by spirometry. Annual rate of change in the FEV1 will be assessed using spirometry. Spirometric measurements are to be performed in triplicate, and the highest value at each time point is to be used for analyses.
Part A and Part B: Plasma Trough Level of Antigenic and Functional A1PI for RYMPHYSIA | Part A, Part B: Pre- and post-dose at multiple timepoints (up to 144 hours) up to Week 104
Part A and Part B: Plasma Concentration of Antigenic and Functional A1PI for RYMPHYSIA | Part A, Part B: Pre- and post-dose at multiple timepoints (up to 144 hours) up to Week 104
Part A and Part B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Part A, Part B: Up to 2 weeks after the last dose (Up to Week 106)
  The number of participants with TEAEs including drug-related AEs, serious AEs (SAEs), and temporally associated AEs will be assessed.
Part A and Part B: Number of Participants Receiving RYMPHYSIA with Development of Post-treatment Immunogenicity as Measured by Anti-A1PI Binding and Neutralizing Antibodies | Part A, Part B: Up to 2 weeks after the last dose (Up to Week 106)
  Serum samples will be analyzed for the presence of antibodies against A1PI using a validated anti-A1PI antibody detection (screening and confirmatory) assay at a qualified specialty laboratory. Samples with confirmed positive titers will be further analyzed for the presence of neutralizing antibodies using a validated neutralizing antibody assay at a qualified specialty laboratory.
Part A and Part B: Changes in Laboratory Assessments | Part A, Part B: Up to 2 weeks after the last dose (Up to Week 106)
  The number of participants who have normal/abnormal values at Baseline compared to normal/abnormal values post-Baseline will be assessed for hematology, clinical chemistry, and urinalysis.
Part A and Part B: Changes in Vital Signs Measurement: Body Temperature | Part A, Part B: Up to 2 weeks after the last dose (Up to Week 106)
  Percent change from Baseline to post Baseline will be assessed for body temperature.
Part A and Part B: Changes in Vital Signs Measurement: Respiratory Rate | Part A, Part B: Up to 2 weeks after the last dose (Up to Week 106)
  Percent change from Baseline to post Baseline will be assessed for respiratory rate.
Part A and Part B: Changes in Vital Signs Measurement: Pulse Rate | Part A, Part B: Up to 2 weeks after the last dose (Up to Week 106)
  Percent change from Baseline to post Baseline will be assessed for pulse rate.
Part A and Part B: Changes in Vital Signs Measurement: Systolic and Diastolic Blood Pressure | Part A, Part B: Up to 2 weeks after the last dose (Up to Week 106)
  Percent change from Baseline to post Baseline will be assessed for systolic and diastolic blood pressure.
Part A and Part B: Number of Participants with Changes in Electrocardiogram (ECG) Measurements | Part A, Part B: Up to 2 weeks after the last dose (Up to Week 106)
Part B: Annual Rate of Change in the Physiologically Adjusted Lung Density | Part B: Up to week 104
  The annual rate of the physiologically adjusted lung density change will be measured as the PD15 of the lung density measurements as assessed by CT densitometry at TLC. CT lung density at the PD15 is the threshold below which 15% of the voxels have lower densities and is used as the parameter for estimating the rate of lung density decline.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/3c7295203e824dad?idFilter=%5B%22TAK-883-4002%22%5D